CLINICAL TRIAL: NCT00296322
Title: A Phase III Randomized Controlled Trial of Adjuvant Chemotherapy for Gastric Adenocarcinoma: Mitomycin and Doxifluridine Versus Intraperitoneal Chemotherapy and Mitomycin, Doxifluridine, and Cisplatin
Brief Title: Trial of Adjuvant Chemotherapy for Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Ulsan University Hospital (Other); Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC0102
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Stomach Cancer
Keywords: stomach cancer; adjuvant chemotherapy; mitomycin; cisplatin; doxifluridine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Mitomycin; doxifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mitomycin-C, Doxifluridine (Active Comparator): Mf: Mitomycin-C 20mg/m2 intravenously (3-6 weeks after surgery) Doxifluridine 460-600mg/m2/day per oral for 3 months (started 4 weeks after surgery)
  Interventions: Drug: cisplatin, mitomycin-C, doxifluridine
- Mitomycin-C, Doxifluridine, Cisplatin (Active Comparator): iceMFP: Cisplatin 100mg with 1L of normal saline intraperitoneally for 2 hours during surgery Mitomycin-C 15mg/m2 intravenously (1 day after surgery) Doxifluridine 460-600mg/m2/day per oral(started at 4 weeks after surgery and administered a total of 12 months) Cisplatin 60mg/m2 intravenously monthly for 6 months (started at 4 weeks after surgery)
  Interventions: Drug: cisplatin, mitomycin-C, doxifluridine

INTERVENTIONS:
Drug: cisplatin, mitomycin-C, doxifluridine — Mf: Mitomycin-C 20mg/m2 intravenously (3-6 weeks after surgery) Doxifluridine 460-600mg/m2/day per oral for 3 months (started 4 weeks after surgery)
  iceMFP: Cisplatin 100mg with 1L of normal saline intraperitoneally for 2 hours during surgery Mitomycin-C 15mg/m2 intravenously (1 day after surgery) Doxifluridine 460-600mg/m2/day per oral(started at 4 weeks after surgery and administered a total of 12 months) Cisplatin 60mg/m2 intravenously monthly for 6 months (started at 4 weeks after surgery)

SUMMARY:
This study is designed to evaluate the efficacy of the intraperitoneal chemotherapy with early mitomycin administration and adding cisplatin to prolonged treatment with doxifluridine compared to mitomycin plus doxifluridine in resected advanced gastric cancer.

DETAILED DESCRIPTION:
Stomach cancer is the most common cancer in Korea and one of the major health problems worldwide. The most effective treatment for gastric cancer is curative surgical resection of primary tumor. However, a substantial number of patients eventually die of recurrences after curative resection. A number of randomized trials investigating the role of adjuvant chemotherapy have been conducted. However, the efficacy of adjuvant chemotherapy is still controversial and varied between Western and Asian trials. Meta-analysis of Western trials didn't demonstrate the benefit of adjuvant chemotherapy after curative resection. Conversely, some Asian studies have demonstrated the efficacy of adjuvant chemotherapy after curative resection. In a previous study, mitomycin plus tegafur prolonged the survival in resected gastric cancer compared to no treatment.

This study is designed to evaluate the efficacy of the intraperitoneal chemotherapy with early mitomycin administration and adding cisplatin to prolonged treatment with doxifluridine compared to mitomycin plus doxifluridine.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven gastric adenocarcinoma
* Grossly serosa invasion of primary tumor is suspicious
* Curative resection was done
* Stage II, IIIA, IIIB, IV (including T4, lesions or N3, but excluding M1 lymph node metastasis)
* Age: 18-69 years old
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2
* Adequate bone marrow function (white blood cell counts ≥ 4,000/ul, platelet count ≥ 100,000/ul, hemoglobin ≥ 10 g/dl)
* Adequate renal function (serum creatinine≤ 1.5)
* Adequate liver function (serum bilirubin ≤1.5 mg/dl, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x normal upper limit)
* Written informed consent was signed by the patient

Exclusion Criteria:

* Previous chemotherapy or radiotherapy
* Active ongoing infection which antibiotic treatment is needed
* Pregnant or lactating women
* Psychosis or convulsion disorder
* Ascites in preoperative abdomen computed tomography (CT)
* Systemic disease which interfere the administration of chemotherapy
* Postoperative pathologic stage IA, IB
* Postoperative pathology indicates that resection margin is involved
* Previous history of other malignancy except cured non-malignant skin cancer and uterine cervical cancer in situ

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2001-10; Primary Completion 2007-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although this study was originally designed to include 528 patients, a total 521 patients could be enrolled.
Groups:
- Mitomycin and Short-term Fluoropyrimidine: Mitomycin-C 20mg/m2 intravenously (3-6 weeks after surgery) Doxifluridine 460-600mg/m2/day per oral for 3 months (started 4 weeks after surgery)
- iceMFP: Intraperitoneal cisplatin, mitomycin, cisplatin and long-term flouropyrimidine
Period: Overall Study
Arm/Group | Mitomycin and Short-term Fluoropyrimidine | iceMFP
Started | 258 | 263
Completed | 237 | 184
Not Completed | 21 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitomycin and Short-term Fluoropyrimidine | iceMFP | Total
Number analyzed (Participants) | 258 | 263 | 521
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 212 | 224 | 436
  >=65 years | 46 | 39 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.87 (10.093) | 52.23 (11.016) | 53.04 (10.591)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 88 | 170
  Male | 176 | 175 | 351
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 258 | 263 | 521

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Mitomycin and Short-term Fluoropyrimidine: Mitomycin and short-term flouropyrimidine
Arm/Group | Mitomycin and Short-term Fluoropyrimidine | iceMFP
Number analyzed (Participants) | 258 | 263
percentage of participants | 50.0 [43.4 to 56.6] | 60.2 [53.6 to 66.7]

2. Secondary Outcome: Toxicity Profile (According to NCI CTC Version 2.0)
Description: Because safety profile in oncology study is evaluated for each toxicity, it is impossible to present the overall patient number. Instead, we presented the number of patients who declined study therapy due to adverse events or patient will.
Time Frame: up to 1 year
Measure: Number; unit: participants
Arm/Group | Mitomycin and Short-term Fluoropyrimidine | iceMFP
Number analyzed (Participants) | 258 | 263
participants | 13 | 30

3. Secondary Outcome: Overall Survival
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mitomycin and Short-term Fluoropyrimidine | iceMFP
Number analyzed (Participants) | 258 | 263
percentage of participants | 59.6 [52.9 to 66.3] | 71.2 [65.1 to 77.3]

ADVERSE EVENTS:
Arm/Group | Mitomycin and Short-term Fluoropyrimidine | iceMFP
Serious Adverse Events (participants affected / at risk) | 0/258 | 0/263
Other Adverse Events (participants affected / at risk) | 230/258 | 251/263
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mitomycin and Short-term Fluoropyrimidine (N=258) | iceMFP (N=263)
Neutropenia (Blood and lymphatic system disorders) | 161 | 217
Anemia (Blood and lymphatic system disorders) | 230 | 238
Thrombocytopenia (Blood and lymphatic system disorders) | 47 | 62
Elevated AST or ALT (Hepatobiliary disorders) | 82 | 60
Hyperbilirubinemia (Hepatobiliary disorders) | 73 | 83
Fatigue (General disorders) | 215 | 236
Anorexia (General disorders) | 203 | 232
Nausea (Gastrointestinal disorders) | 187 | 226
Vomiting (Gastrointestinal disorders) | 73 | 126
Stomatitis (Gastrointestinal disorders) | 55 | 114
Constipation (Gastrointestinal disorders) | 85 | 164
Diarrhea (Gastrointestinal disorders) | 168 | 193
Alopecia (General disorders) | 139 | 212
Neuropathy (Nervous system disorders) | 46 | 165
Myalgia (Musculoskeletal and connective tissue disorders) | 54 | 91
Edema (Musculoskeletal and connective tissue disorders) | 20 | 74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No